CLINICAL TRIAL: NCT02215434
Title: Phase 2 Study of Transdermal Testosterone for Low Libido in Pre and Postmenopausal Women
Brief Title: Safety Study of Transdermal Testosterone for Low Libido in Pre and Postmenopausal Women
Acronym: TESTOSTERONE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Potiguar (Other)
Collaborators: Universidade Federal do Ceara (Other); Federal Institute of Science and Technology of Ceara (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UNP/CNPq02
Record Dates: First submitted 2014-08-12; First posted 2014-08-13 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Sex Behavior
Keywords: Libido; Sexual Dysfunction; testosterone
MeSH Terms: conditions — Sexual Behavior; Sexual Dysfunction, Physiological | interventions — Testosterone; Administration, Cutaneous

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Biolipid B2 (blanked/placebo) (Placebo Comparator): The study is a single-center, single-blind, placebo-controlled, parallel group trial.
  It consists of a 4-week screening period plus a 12-week treatment phase. At the screening visit, all participants underwent a physical examination including vital signs and breast and pelvic examination.
  They were randomly assigned in a 1:1 ratio to receive a transdermal vehicle biolipid B2 (identical placebo) provided by Evidence Pharmaceuticals Inc, SP,BRAZIL.
  The testosterone and placebo emulsion were alcohol-free matrixes that were applied topically to the forearm daily for the period of 12 weeks.
  Interventions: Drug: Biolipid B2 (blanked/placebo); Drug: Testosterone, Transdermal, Behavior
- Testosterone, Transdermal, Behavior (Active Comparator): Testosterone 0.5%, daily, 3 months
  Interventions: Drug: Biolipid B2 (blanked/placebo); Drug: Testosterone, Transdermal, Behavior

INTERVENTIONS:
Drug: Biolipid B2 (blanked/placebo) — the intervention will be the comparison effects of both emulsions
  Other Names: Biolipid B2 0.5% testosterone, Evidence, Fortaleza, Brazil; Biolipid B2 0.5% testosterone, Pharmacom, São Paulo, Brazil
Drug: Testosterone, Transdermal, Behavior — Transdermal 0.5% testosterone Biolipid/B2
  Other Names: Transdermal testosterone Biolipid/B2

SUMMARY:
Female sexual dysfunction (FSD) is an established side effect of Selective serotonin reuptake inhibitors (SSRIs) and serotonin noradrenalin reuptake inhibitors (SNRIs), causing symptoms such as loss of libido, arousal difficulties, or delayed orgasm or anorgasmia.

Efficacy of testosterone therapy for the treatment of hypoactive sexual desire disorder (HSDD) in women has been demonstrated in studies including naturally and surgically menopausal women, either alone or in combination with estrogen, with or without progestin therapy.

DETAILED DESCRIPTION:
Recent studies have reported an increase in the number of satisfactory sexual events recorded in a 4-week daily diary, as a primary outcome, and reduction in associated personal distress.

There is also evidence that testosterone therapy results in a similar improvement in sexual function in premenopausal women with loss of libido.

Testosterone therapy has been associated with significantly improved well-being in studies in which the participants had low well-being at enrollment.

Trials of testosterone for HSDD in women have excluded those with clinical depression, as well as those taking antidepressants.

Whether testosterone will benefit women with HSDD who are taking an antidepressant is not known.

The primary aim of this study was to examine the effects of transdermal testosterone therapy with a nanoemulsion BIOLIPID B2 on sexual function in women at midlife, who were experiencing treatment-emergent low libido. The primary study outcome was the change in the total score of the Sabbatsberg Sexual Self-rating Scale (SSS).

In line with previous studies of women without depression, efficacy was measured by the change in the frequency of SSEs over 4 weeks, as well as the domains of the SSS, general well-being, depression, and mood status.

In this present study these factors will be analized in 12 weeks interval

ELIGIBILITY:
Inclusion Criteria:

* a body mass index between 18 and 35 kg/m2
* diminished libido complaints
* no evidence of severe clinical depression
* participants in good health based on history and physical examination.

Exclusion Criteria:

* a past history of neurological disorder
* recent psychiatric or systemic illness
* use of psychoactive medications
* alcohol excess consumption or any other drug abuse.
* women who had under gone treatment for cardiovascular disease, genital bleeding, acne, depression, dyspareunia or those who had received oral androgen therapy in the previous 3 months were excluded
* in addition women taking medications known to interfere with sex steroid metabolism were also excluded.

Ages: 18 Years to 89 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-09; Primary Completion 2013-04 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
satisfactory sexual events | 12 weeks
  Recent studies have reported an increase in the number of satisfactory sexual events (SSEs) recorded in a 4-week daily diary, as a primary outcome, and reduction in associated personal distress.

SECONDARY OUTCOMES:
Total testosterone and SHBG levels at screening and after 12 weeks of treatment. | 12 weeks
  Total testosterone and SHBG levels were determined at screening and week 12.

OTHER OUTCOMES:
Safety of transdermal Testosterone Biolipid B2 effects | 12 weeks
  Safety is assessed by comparing the rates of adverse events in the two treatment groups. Androgenic side effects including the frequency of facial depilation per month, hirsutism by the Ferriman-Gallwey scale (range 0-4 for each of nine body regions), acne by the Palatsi scale and clitoromegaly by examination were assessed at screening and the final visit.
  We also monitor vital signs and concomitant medications.

CONTACTS AND LOCATIONS:
Overall Officials: MARCO A BOTELHO, M.Sc., Ph.D, Study Director — University Potiguar; Dinalva B Queiroz, PhD, Principal Investigator — University Potiguar
Locations (1):
- University Potiguar, Natal, Rio Grande do Norte, Brazil

REFERENCES:
- [Result] Botelho MA, Queiroz DB, Barros G, Guerreiro S, Fechine P, Umbelino S, Lyra A, Borges B, Freitas A, Queiroz DC, Ruela R, Almeida JG, Quintans L Jr. Nanostructured transdermal hormone replacement therapy for relieving menopausal symptoms: a confocal Raman spectroscopy study. Clinics (Sao Paulo). 2014 Feb;69(2):75-82. doi: 10.6061/clinics/2014(02)01. PMID 24519196
- See also: Article — http://www.scielo.br/scielo.php?script=sci_arttext&pid=S1807-59322014000200075&lng=en&nrm=iso&tlng=en